CLINICAL TRIAL: NCT06186323
Title: Examining the Relationship Between Opportunities Offered in the Home Environment and Motor Development and Sensory Processing in Children Diagnosed With Congenital Muscular Torticollis
Brief Title: Relationship Between Home Environment and Development in Children Diagnosed With Muscular Torticollis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Rabia ZORLULAR, principal investigator, Gazi University
Other Study IDs: Torticollis and affordance
Record Dates: First submitted 2023-12-15; First posted 2024-01-02 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Congenital Muscular Torticollis; Motor Development; Sensory Integration Disorder
Keywords: Torticollis; Motor development; Sensory Integration; Home environment
MeSH Terms: conditions — Congenital torticollis; Torticollis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- congenital muscular torticollis: 40 children diagnosed with congenital muscular torticollis, aged 0-15 months, with parental consent, without any vision or hearing problems, will be included in the study. Children with chromosomal anomalies, serious congenital problems and whose parents do not volunteer to participate will not be included in the study.
  During the evaluations, the demographic characteristics of the babies (gender, gestational age, birth weight, parental information, mother's pregnancy type, pregnancy history, Apgar score) will be recorded from the file and by interviewing the family. Photographs will be taken to ensure an objective evaluation. The Affordances in the Home Environment for Motor Development-Infant Scale will be used to explore and evaluate the home environment. It was planned to use the Test of Sensory Functions in Infants to evaluate the sensory development of babies. It is planned to use Peabody Motor Development Scale-2 to evaluate motor development.
  Interventions: Behavioral: Affordances in the Home Environment for Motor Development-Infant Scale; Behavioral: Peabody Developmental Motor Scales-2; Behavioral: Test Of Sensory Functions In Infants (TSFI)

INTERVENTIONS:
Behavioral: Affordances in the Home Environment for Motor Development-Infant Scale — Affordances in the Home Environment for Motor Development-Infant Scale is a parent-filled assessment to determine the nature and amount of factors affecting infant motor skill development in the home environment, including the availability of toys, materials, and the availability of spaces.
Behavioral: Peabody Developmental Motor Scales-2 — Peabody Developmental Motor Scales | Second Edition (PDMS-2) combines in-depth assessment with training or remediation of gross and fine motor skills of children from birth through 5 years. Used to evaluate children's motor development with separate tests and rating scales for both gross motor skills and fine motor skills
Behavioral: Test Of Sensory Functions In Infants (TSFI) — his test helps you identify infants with sensory integrative dysfunction-including those at risk for developing learning disabilities as they grow older. The TSFI provides objective criteria that allow you to determine whether, and to what extent, an infant has deficits in sensory functioning. Designed for use with children from 4 months to 18 months old, the TSFI provides an overall measure of sensory processing and reactivity, as well as scores on the following subdomains: Reactivity to Tactile Deep Pressure Visual Tactile Integration Adaptive Motor Function Ocular Motor Control Reactivity to Vestibular Stimulation

SUMMARY:
Congenital muscular torticollis (CMT) is a common postural deformity that occurs shortly after birth and is typically characterized by ipsilateral cervical lateral flexion and contralateral cervical rotation due to unilateral shortening of the sternocleidomastoid (SKM) muscle. It is a non-neurological postural disorder that generally affects 3% to 16% of babies. Theories such as intrauterine stenosis, vascular causes, fibrosis of the peripartum bleeding area, difficult birth, and primary myopathy of the SCM muscle have been put forward for its causes.Head position; It is thought that it may cause a negative impact on posture control and movement development, sensorimotor coordination, and retardation in gross motor function by affecting the shoulder, rib cage and abdominal muscles. Motor skills and sensory experiences begin to develop after birth and development continues as children grow. Having good motor control also helps children explore the world around them, which can help many other areas of development. There are many environmental and biological factors that affect motor development. In particular, the home environment, where the child spends most of his time, is one of the key factors affecting motor development. The home environment is known to be a very important factor for motor development in babies. At the same time, the variety of equipment and environmental conditions help children provide different sensory experiences. Since it is a common practice for physiotherapists to advise patients on home activities, exploring the home environment can have important effects on development. For these reasons, it was thought that the motor development and sensory processing suggestions given in the home environment for children diagnosed with torticollis would be supported by home environment opportunities.

DETAILED DESCRIPTION:
It is thought that Congenital muscular torticollis (CMT) affects the muscles as well as the development of the head and face, causing various asymmetries, delays in gross motor functions, and disorders in posture and balance control. Bent neck position can cause plagiocephaly. Characteristic craniofacial deformities are asymmetry in the eyebrows and cheekbones, deviation of the chin and nose tip, inferior orbital abnormality on the affected side, asymmetry in ear placement, and shortening of the vertical dimension of the ipsilateral face. It has been shown that in later periods, it may cause asymmetry in the use of the upper extremities in children, delay in gross motor functions, and effects on posture and balance control. Head position; It is thought that it may cause a negative impact on posture control and movement development, sensorimotor coordination, and retardation in gross motor function by affecting the shoulder, rib cage and abdominal muscles. Motor skills and sensory experiences begin to develop after birth and development continues as children grow. Having good motor control also helps children explore the world around them, which can help many other areas of development. There are many environmental and biological factors that affect motor development. Especially the home environment, where the child spends most of his time, is one of the key factors affecting motor development. The home environment is known to be a very important factor for motor development in babies. At the same time, the variety of equipment and environmental conditions help children provide different sensory experiences. Since it is a common practice for physiotherapists to advise patients on home activities, exploring the home environment can have important effects on development. For these reasons, it was thought that the motor development and sensory processing suggestions given in the home environment for children diagnosed with torticollis would be supported by home environment opportunities. This study was planned to examine the relationship between the opportunities offered in the home environment and motor development and sensory processing in children diagnosed with congenital muscular torticollis.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-15 months, with parental consent,
* Diagnosed with congenital muscular torticollis
* Their families will be included.

Exclusion Criteria:

* Children with chromosomal anomalies,
* serious congenital problems
* those whose parents do not volunteer to participate will not be included in the study.

Ages: 1 Month to 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 40 children diagnosed with congenital muscular torticollis, aged 0-15 months, with parental consent, without any vision or hearing problems, will be included in the study. severe chromosomal abnormality Children with congenital problems and whose parents do not volunteer to participate will not be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Affordances in the Home Environment for Motor Development-Infant Scale | 1-15 months
  Affordances in the Home Environment for Motor Development-Infant Scale is a parent-filled assessment to determine the nature and amount of factors affecting infant motor skill development in the home environment, including the availability of toys, materials, and the availability of spaces. The scale consists of 41 items in total. For babies aged 3-12 months, questions up to the first 32 items are answered. It is stated that other substances are not suitable for babies under 12 months. All substances are applied to babies between 12-18 months. Questions answered as yes or no are scored as 0.1 (0: no, 1: yes). Other questions are scored as 0, 1, 2, 3. For babies up to 12 months, a total of 66 points is obtained. For babies older than 12 months, a total of 93 points is obtained. A higher score indicates better environmental enrichment.
Peabody Developmental Motor Scales | Second Edition | 1-15 months
  Peabody Developmental Motor Scales | Second Edition (PDMS-2) combines in-depth assessment with training or remediation of gross and fine motor skills of children from birth through 5 years. It consists of gross motor and fine motor parts. The Gross motor section includes 151 items from 4 subtests: reflexes, stasis, locomotion, and object manipulation. The fine motor section consists of 2 subtests and 98 items: comprehension and visual-motor integration. The total motor part is the sum of the items in the gross and fine 25 motor parts. Items are scored with 0, 1, and 2 points. When the child performs the item according to the specified item criteria, 2 points are given. 1 point is awarded when the behavior occurs but the criteria for successful performance are not fully met. A score of 0 is given when the child is unable to try the item or does not reveal any skills when he tries it. Results are expressed as a raw score, standard score, or total motor score.
Test of Sensory Functıons ın Infants | 1-15 months
  It was planned to useTest of Sensory Functıons ın Infants (TSFI) to evaluate the sensory development of babies. BDFT is frequently used to evaluate the sensory processing functions of babies aged 4-18 months. It is used to determine whether a baby has a sensory processing problem and to what extent. It consists of 24 items.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia ERASLAN, Principal Investigator — Study Principal Investigator-Gazi University
Locations (1):
- Rabia ERASLAN, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ohman A, Nilsson S, Lagerkvist AL, Beckung E. Are infants with torticollis at risk of a delay in early motor milestones compared with a control group of healthy infants? Dev Med Child Neurol. 2009 Jul;51(7):545-50. doi: 10.1111/j.1469-8749.2008.03195.x. Epub 2009 Jan 26. PMID 19191832
- [Result] Sargent B, Kaplan SL, Coulter C, Baker C. Congenital Muscular Torticollis: Bridging the Gap Between Research and Clinical Practice. Pediatrics. 2019 Aug;144(2):e20190582. doi: 10.1542/peds.2019-0582. PMID 31350358
- [Result] Cacola PM, Gabbard C, Montebelo MI, Santos DC. Further Development and Validation of the Affordances in the Home Environment for Motor Development-Infant Scale (AHEMD-IS). Phys Ther. 2015 Jun;95(6):901-23. doi: 10.2522/ptj.20140011. Epub 2014 Dec 18. PMID 25524875
- [Result] Chiarello LA, Palisano RJ. Investigation of the effects of a model of physical therapy on mother-child interactions and the motor behaviors of children with motor delay. Phys Ther. 1998 Feb;78(2):180-94. doi: 10.1093/ptj/78.2.180. PMID 9474110